CLINICAL TRIAL: NCT03389815
Title: The Dose-escalation Study Followed by an Extension Phase Evaluating the Safety, Pharmacokinetics and Efficacy of WX-0593 in Advanced Solid Tumor Patients With Anaplastic Lymphoma Kinase（ALK）/Receptor Tyrosine Kinase（ROS1） Positive
Brief Title: A Study Evaluates the Safety, Pharmacokinetics and Efficacy of WX-0593 in Advanced Solid Tumor Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WX0593-001
Record Dates: First submitted 2017-12-06; First posted 2018-01-04 (Actual); Last update posted 2018-01-04 (Actual); Status verified 2017-12

CONDITIONS: Advanced Solid Tumor, Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WX-0593 Tablets (Experimental): The first part is a dose-escalation design in patients with ALK/ROS1-positive solid tumor. The second part is an expansion in non-small cell lung Cancer (NSCLC) characterized by abnormalities in ALK expression.
  Interventions: Drug: WX-0593 Tablets

INTERVENTIONS:
Drug: WX-0593 Tablets — tablets, dosage ranged from 30 mg to 300 mg, quaque die（QD）
  Other Names: FL-006

SUMMARY:
The purpose of the study is to evaluate safety, pharmacokinetics and efficacy of WX-0593 alone in the treatment of advanced cancer.

DETAILED DESCRIPTION:
The first part is a single-arm, phase 1, open label, dose-escalation design in patients with anaplastic lymphoma kinase（ALK）/receptor tyrosine kinase（ROS1） Positive ALK/ROS1-positive solid tumor. The second part is an expansion in non-small cell lung Cancer (NSCLC) characterized by abnormalities in anaplastic lymphoma kinase(ALK) expression.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 70 years, inclusive.
2. Female or male
3. Patient has an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1.
4. Life expectancy of at least 12 weeks.
5. At least one measurable lesion (according to RECIST v1.1)
6. Histologically or cytologically confirmed diagnosis of advanced solid tumor malignancy with ALK/ROS1+ (For the expansion phase, patients must have NSCLC with ALK+ ):

   * Patients with advanced tumor (eg. NSCLC, lymphoma, inflammatory myofibroblastic tumor) who failed in standard treatment (eg. resistant of ALK inhibitors or chemotherapy)
   * Patients with advanced NSCLC who cannot accept chemotherapy or intolerance with chemotherapy.
   * Advanced NSCLC patients who could not afford ALK inhibitor treatment.
7. Patients with treated or untreated asymptomatic Central Nervous System（CNS） metastases may be allowed to enroll.
8. Patients must have normal function as defined: ANC≥1.5*10^9/L PLT≥100*10^9/L， Total Bilirubin （TBIL）≤1.5*Upper Limit of Normal（ULN） ( Gilbert's Syndrome TBIL ≤3.0*ULN and DBIL≤1.5*ULN )，Alanine Transaminase （ALT）and Aspartate Aminotransferase（AST）≤2.5*ULN. For liver metastasis patients, ALT and AST≤5*ULN, Cr≤1.5*ULN, LVEF≥50%.
9. Any surgery or radiation (expect for palliative radiation) must have been completed at least 4 weeks prior to first dosing. Palliative radiation must have been completed at least 48 hours prior to first dosing.
10. All related adverse events from previous anti-cancer therapies must have recovered to ≤ Grade 1 (except for alopecia).
11. Patients must be able to understand and volunteer to sign the informed consent.

Exclusion Criteria:

1. Clinically significant cardiovascular disease within 3 months prior to first dosing.
2. Ongoing cardiac dysrhythmias, or any grade of uncontrolled atrial fibrillation, or prolonged QT interval (QTc > 480 ms).
3. Patients need medications that may prolong QT interval or induce torsades de pointes within 14 days prior to the first dosing or during the study.
4. Peripheral neuropathy ≥ Grade 3 according to CTCAE 4.03.
5. Patients who received continuous use of steroids for more than 30 days, or who need long-term use of steroid hormones or other immunosuppressive agents.
6. History of extensive disseminated/bilateral pulmonary interstitial fibrosis, interstitial fibrosis or interstitial lung disease of Grade 3/4 .
7. Presence of active gastrointestinal (GI) disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of WX-0593.
8. Patients who are receiving warfarin sodium (Coumadin) or any other coumadin-derived anticoagulants，and patients with coagulation disturbance and bleeding tendency.
9. Patient has received other investigational drug within 1 month.
10. Patients with acute or chronic infectious medical conditions, including active hepatitis (Hepatitis A、 Hepatitis B、 Hepatitis C ) or HIV infection.
11. Patients who received prior anti-cancer therapy within 2 weeks (t1/2 ≤ 3 days) or within 4 weeks (3 days < t1/2）. Patients previously treated with crizotinib could start WX-0593 dosing after 1 week from the last dosing.
12. Patients who could not discontinue therapy with potent CYP3A4 inhibitors or inducers within 1 week prior first dosing, or patients who need therapy with CYP3A4 inhibitors or inducers during the study.
13. Patients received medications known to be metabolized by CYP3A4 and with narrow therapeutic indices, who could not discontinue within 1 week prior to the start of WX-0593 administration. Patients who need therapy with those medications during the study.
14. Females who are pregnant or breastfeeding.
15. Patients with childbearing potential must agree to use adequate contraception for the duration of treatment and for 6 months after the study.
16. Drug abusers and alcoholics.
17. History of definite nerves or psychosis diseases including epilepsy or dementia.
18. History of other malignancy.
19. Concurrent condition that in the investigator's opinion would jeopardize compliance with the protocol or would impart excessive risk associated with study participation that would make it inappropriate for the patient to be enrolled.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2017-09-14 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose（MTD） | 28 days
  The MTD is determined by the number of the participants in cohort who suffer a dose-limiting toxicity (DLT). The MTD is defined as the former dose at which more than one third of the participants develop a DLT. If no DLTs are observed, the MTD is not reached.

SECONDARY OUTCOMES:
Tmax of WX-0593 | 28 days
  Pharmacokinetics of WX-0593 by assessment of time to Cmax
Cmax of WX-0593 | 28 days
  Pharmacokinetics of WX-0593 by assessment of maximum plasma WX-0593 concentration.
Cmin of WX-0593 | 28 days
  Pharmacokinetics of WX-0593 by assessment of minimum plasma WX-0593 concentration.
AUC of WX-0593 | 28 days
  Pharmacokinetics of WX-0593 by assessment of area under the plasma concentration time curve from zero to infinity
tl/2 of WX-0593 | 28 days
  Pharmacokinetics of WX-0593 by assessment of the terminal half-life
Cssmin of WX-0593 | 28 days
  Cmin of WX-0593 at steady state
Cssmax of WX-0593 | 28 days
  Cmax of WX-0593 at steady state
Css-av of WX-0593 | 28 days
  Mean plasma concentration of WX-0593 at steady state
AUCss of WX-0593 | 28 days
  area under the curve of WX-0593 at steady state
DF of WX-0593 | 28 days
  Pharmacokinetics of WX-0593 by assessment of degree of fluctuation
Vz of WX-0593 | 28 days
  volume of distribution during terminal phase after WX-0593 administration
CLs of WX-0593 | 28 days
  total plasma,serum or blood clearance of WX-0593 after administration
Objective Response Rate (ORR) | From fist administration of WX-0593 to 28 days after last medication.
  Primary efficacy endpoint is a change in the proportion of subjects showing overall objective response rate (ORR) from baseline to final tumor assessment point after treatment. As Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria, the percentage of subjects indicating PR (partial response) and CR (complete response) will be calculated.
  According to RECIST 1.1 criteria, complete response (CR) - the disappearance of all target lesions and partial response ( PR ) - at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum of longest diameter.
Progression-free survival (PFS) | From fist administration of WX-0593 to 28 days after last medication.
  PFS defined as the time from baseline to first observed disease progression or death from any cause.
Disease Control Rate (DCR) | From fist administration of WX-0593 to 28 days after last medication.
  DCR is the percentage of patients with best response of CR, PR or Stable Disease (SD).
  SD was defined as neither sufficient shrinkage to qualify for a PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of the longest diameter.
Duration of Response (DOR) and so on | From fist administration of WX-0593 to 28 days after last medication.
  The DOR is defined as the time from the date of the first response CR/PR (whichever is first recorded) to the date on which progressive disease (PD) is first noted or date of death.

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, M.D., Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Jian Fang, M.D., Principal Investigator — Peking University Cancer Hospital & Institute; Shucai Zhang, M.D., Principal Investigator — Beijing Chest Hospital, Capital Medical University; Yunpeng Liu, M.D., Principal Investigator — First Hospital of China Medical University
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang G, Wang Y, Zhao H, Zheng Q, Wang X, Jia L, Xin Q, Ma C, Zhang Y, Zheng S, Kang X. Translational Model-Informed Dose Selection for Iruplinalkib, a Selective Oral ALK/ROS1 Tyrosine Kinase Inhibitor. Clin Transl Sci. 2025 Jul;18(7):e70287. doi: 10.1111/cts.70287. PMID 40650620
- [Derived] Shi Y, Fang J, Hao X, Zhang S, Liu Y, Wang L, Chen J, Hu Y, Hang X, Li J, Liu C, Zhang Y, Wang Z, Hu Y, Gu K, Huang J, Zhang L, Shan J, Ouyang W, Zhao Y, Zhuang W, Yu Y, Zhao J, Zhang H, Lu P, Li W, Si M, Ge M, Geng H. Safety and activity of WX-0593 (Iruplinalkib) in patients with ALK- or ROS1-rearranged advanced non-small cell lung cancer: a phase 1 dose-escalation and dose-expansion trial. Signal Transduct Target Ther. 2022 Jan 28;7(1):25. doi: 10.1038/s41392-021-00841-8. PMID 35087031